CLINICAL TRIAL: NCT02756845
Title: A Phase 1, Multi-center, Open-label, Dose De-escalation Study to Evaluate the Safety and Efficacy of Talimogene Laherparepvec in Pediatric Subjects With Advanced Non Central Nervous System Tumors That Are Amenable to Direct Injection
Brief Title: Study of Talimogene Laherparepvec In Children With Advanced Non CNS Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20110261; 2015-003645-25 (EudraCT Number)
Record Dates: First submitted 2015-12-15; First posted 2016-04-29 (Estimated); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Advanced Non CNS Tumors
Keywords: Non CNS Tumor
MeSH Terms: interventions — talimogene laherparepvec

STUDY DESIGN:
Intervention Model Description: Approximately 18 to 24 treated pediatric subjects are expected to be enrolled into 2 cohorts stratified by age (permissible based on the incidence of DLTs, a minimum of 6 subjects/cohort and a minimum of 18 subjects total).
  * Cohort A1 (12 to ≤ 21 years of age)
  * Cohort B1 (2 to < 12 years of age) Initially, 3 subjects 12 to ≤ 21 years of age are to be enrolled and treated at 100% of the recommended adult dose regimen of talimogene laherparepvec (cohort A1). The dose level review team (DLRT) will review the safety data of the first 3 subjects in the older age cohort A1 to decide if the younger age cohort B1 can be opened for enrollment. If a DLT occurs in the first 3 DLT-evaluable subjects in the older age cohort (A1 or A2), the younger age cohort will not open until a DLT rate < 33% is observed with at least 6 DLT-evaluable subjects in the older age cohort (A1 or A2).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Talimogene Laherparepvec (TVEC) (Experimental): The first dose of talimogene laherparepvec will be administered at a dose of up to 4.0 mL of 10ᶺ6 PFU/mL followed by a dose of up to 4.0 mL of 10ᶺ8 PFU/mL 21 days (+3 days) later. Subsequent doses of up to 4.0 mL of 10ᶺ8 PFU/mL will be administered every 14 days (± 3 days) thereafter. Cohorts will be assigned as follows: Cohort A1 (age 12 to ≤ 21 years). Cohort B1 (age 2 to < 12 years). The DLRT will review the safety data of the first 3 subjects in the older age cohort A1 to decide if the younger age cohort B1 can be opened for enrollment. If dose de-escalation is needed and if permissible based on the incidence of DLTs, additional DLT-evaluable subjects will be enrolled and treated at a lower dose level of talimogene laherparepvec. Dose de-escalation cohorts will be assigned as follows and the same DLT rules will be applied: Cohort A2 (age 12 to ≤ 21 years), Cohort B2 (age 2 to < 12 years).
  Interventions: Drug: Talimogene Laherparepvec

INTERVENTIONS:
Drug: Talimogene Laherparepvec — Talimogene laherparepvec will be administered by intralesional injection only into injectable cutaneous, subcutaneous, nodal tumors, and other non-visceral tumors with or without image ultrasound guidance. The first dose of talimogene laherparepvec will be up to 4.0 mL of 10^6 PFU/mL administered on day 1. The second injection, up to 4.0 mL of 10^8 PFU/mL (or up to 4.0 mL of 10^6 PFU/mL for a dose de-escalated cohort), will be administered 21 (+3) days after the initial injection. All subsequent injections, up to 4.0 mL of 10^8 PFU/mL (or up to 4.0 mL of 10^6 PFU/mL for a dose de-escalated cohort), will be administered every 14 (± 3) days. The treatment cycle interval may be increased due to toxicity.
  Other Names: TVEC

SUMMARY:
This is a phase 1 study to evaluate the safety of intralesional talimogene laherparepvec administration in pediatric subjects with advanced non-CNS tumors that are amenable to direct injection

DETAILED DESCRIPTION:
This is a phase 1, multicenter, open-label study of talimogene laherparepvec in pediatric subjects with advanced non-CNS tumors that are amenable to direct injection in the clinical setting. Approximately 18 - 24 pediatric subjects are expected to be enrolled and treated with at least 1 dose of talimogene laherparepvec into 2 cohorts stratified by age. DLT will be evaluated based on at least 9 DLT-evaluable subjects in cohort A1. The DLT evaluation period is 35 days from the initial administration of talimogene laherparepvec.

ELIGIBILITY:
Inclusion Criteria

* Subject's legally acceptable representative has provided informed consent/assent when the subject is legally too young to provide informed consent/assent and the subject has provided written assent based on local regulations and/or guidelines prior to any study-specific activities/procedures being initiated.
* Should be willing to submit local HSV-1 serostatus within 28 days prior to enrollment.
* Subject must be a candidate for intralesional injection, defined as one or more of the following:

  * at least 1 injectable lesion ≥ 10 mm in longest diameter
  * multiple injectable lesions that in aggregate have a longest diameter of ≥ 10 mm
* Life expectancy > 4 months from the date of enrollment.
* Male or female subjects 2 to ≤ 21 years of age at the time of informed consent/assent.
* Histologically or cytologically confirmed non-CNS solid tumor that recurred after standard/frontline therapy, or for which there is no standard/frontline therapy available.
* Presence of measurable or non-measurable lesions as defined by irRC-RECIST
* Performance status as per protocol
* Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to dosing.
* Adequate organ function as defined in protocol

  •Exclusion Criteria
* Diagnosis of leukemia, non-Hodgkin's lymphoma, Hodgkin's disease, or other hematologic malignancy.
* Radiotherapy to the bone marrow within 6 weeks prior to enrollment OR within 3 months prior to enrollment if prior radiotherapy to the craniospinal axis or to at least 60% of the pelvis was received; within 2 weeks prior to enrollment if local palliative radiotherapy was received.
* Primary ocular or mucosal melanoma.
* History of other malignancy within the past 5 years with the following exception:

  • malignancy treated with curative intent and with no known active disease present and has not received chemotherapy for > 5 years before enrolment and felt to be at low risk for recurrence by the treating physician.
* History or evidence of active autoimmune disease that requires systemic treatment (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Active herpetic skin lesions or prior complications of herpetic infection (eg, herpetic keratitis or encephalitis).
* Prior treatment with talimogene laherparepvec or any other oncolytic virus.
* Prior treatment with a tumor vaccine.
* Requires intermittent or chronic treatment with an antiherpetic drug (eg, acyclovir), other than intermittent topical use.
* Expected to require other cancer therapy while on study with the exception of local palliative radiation treatment.
* Has acute or chronic active hepatitis B virus or hepatitis C virus infection or received treatment with nucleotide analogs such as those used in the treatment of hepatitis B virus (eg, lamivudine, adefovir, tenofovir, telbivudine, and entecavir), ribavirin, or interferon alpha within 12 weeks of initiation of study treatment.
* Known or suspected human immunodeficiency virus (HIV) infection.
* Received live vaccine within 28 days prior to enrollment.
* No antiplatelet or anticoagulation medications allowed within 7 days prior totalimogene laherparepvec injection except low-dose heparin needed to maintain venous catheter patency.
* Female subject is pregnant or breast-feeding, or planning to become pregnant during study treatment and through 3 months after the last dose of talimogene laherparepvec.
* Female subject of childbearing potential who is unwilling to use acceptable method(s) of effective contraception during study treatment and through 3 months after the last dose of talimogene laherparepvec. Note: Acceptable methods of effective contraception are defined in the informed consent/assent form. Where required by local laws and regulations, additional country-specific contraception requirements may be outlined in a country-specific protocol supplement at the end of the Appendix Section of protocol.
* Subject has known sensitivity to any of the products or components to be administered during dosing.
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the subject and investigator's knowledge.
* History or evidence of any psychiatric disorder, substance abuse or any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
* Subject who is unwilling to minimize exposure with his/her blood or other body fluids to individuals who are at higher risks for HSV-1 induced complications (immunosuppressed individuals, HIV-positive individuals, pregnant women, or children under the age of 1 year) during talimogene laherparepvec treatment and through 28 days after the last dose of talimogene laherparepvec.
* Evidence of clinically significant immunosuppression such as the following:

  * primary immunodeficiency state such as severe combined immunodeficiency disease
  * concurrent opportunistic infection
  * receiving systemic immunosuppressive therapy (> 2 weeks prior to enrollment), including oral steroid doses (with the exception of maintenance physiologic replacement). Subjects who require intermittent use of steroids for inhalation or local steroid injection will not be excluded from the study
  * less than 6 months from autologous bone marrow transplant or stem cell infusion
  * history of allogeneic bone marrow transplant
* History or evidence of xeroderma pigmentosum.
* Sexually active subjects and their partners unwilling to use a male or female latex condom to avoid potential viral transmission during sexual contact while on treatment and within 30 days after treatment with talimogene laherparepvec. For those with latex allergies, polyurethane condoms may be used.
* Prior chemotherapy, treatment dose radiotherapy, or biological cancer therapy within 14 days prior to enrollment or has not recovered to Common Terminology Criteria for Adverse Events version 4.0 (CTCAE) grade 1 or better from adverse event due to cancer therapy administered more than 14 days prior to enrollment.
* CNS tumor or clinically active brain metastases (patient with a history of treated brain metastases are eligible if there is radiographic evidence of improvement upon the completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study).
* Currently receiving treatment in another investigational device or drug study, or less than 14 days since ending treatment on another investigational device or drug study(ies) or has not recovered to CTCAE version 4.0 grade 1 or better from adverse event due to other investigational device or drug study administered more than 14 days prior to enrollment. Other investigational procedures while participating in this study are excluded.
* Major surgery ≤ 14 days prior to enrollment or has not recovered to CTCAE version 4.0 grade 1 or better from adverse event due to surgery performed more than 14 days prior to enrollment.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (22):
- United States (9):
  - AI Dupont Hospital for Children, Wilmington, Delaware
  - Nemours du Pont Hospital in Florida, Jacksonville, Florida
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Childrens Hospital of Michigan, Detroit, Michigan
  - Columbia University Medical Center, New York, New York
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Childrens Hospital, Columbus, Ohio
  - Childrens Hospital of Philidelphia, Philadelphia, Pennsylvania
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Centre Hospitalier Universitaire Sainte Justine, Montreal, Quebec, Canada
- France (3):
  - Institut Hematologie et Oncologie Pediatrique, Lyon
  - Centre Hospitalier Universitaire de Marseille - Hopital de la Timone, Marseille
  - Institut Curie, Paris
- IRCCS Ospedale Pediatrico Bambino, Roma, Italy
- Spain (5):
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Catalonia
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
  - Hospital Universitario Infantil Niño Jesus, Madrid
- Switzerland (2):
  - Universitaets-Kinderspital beider Basel, Basel
  - Universitaets-Kinderspital, Zurich

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Moreno L, Teira P, Croop JM, Gerber NU, Andre N, Aerts I, Gros Subias L, De Wilde B, Bautista F, Turpin B, Kunduri S, Hamidi A, Lawrence T, Streby KA. A phase 1, first-in-child, multicenter study to evaluate the safety and efficacy of the oncolytic herpes virus talimogene laherparepvec in pediatric patients with advanced solid tumors. Front Pediatr. 2023 May 24;11:1183295. doi: 10.3389/fped.2023.1183295. eCollection 2023. PMID 37292376
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 15 participants were enrolled across 11 centers in Belgium, Canada, France, Spain, Switzerland and the United States from August 2017 to November 2022.
Groups:
- Cohort A1: Talimogene Laherparepvec (TVEC) - Aged 12 to ≤ 21 Years: Participants aged 12 to ≤ 21 years were administered an initial dose of talimogene laherparepvec at a dose of up to 4.0 mL of 10ᶺ6 PFU/mL followed by a dose of up to 4.0 mL of 10ᶺ8 PFU/mL 21 days (± 3) later. All subsequent injections, up to 4.0 mL of 10^8 PFU/mL were administered every 14 (± 3) days for up to approximately 9 months. Talimogene laherparepvec was administered by intralesional injection only into injectable cutaneous, subcutaneous, nodal tumors, and other non-visceral tumors with or without image ultrasound guidance.
- Cohort B1: Talimogene Laherparepvec (TVEC) - Aged 2 to < 12 Years: Participants aged 2 to < 12 years were administered an initial dose of talimogene laherparepvec at a dose of up to 4.0 mL of 10ᶺ6 PFU/mL followed by a dose of up to 4.0 mL of 10ᶺ8 PFU/mL 21 days (± 3) later. All subsequent injections, up to 4.0 mL of 10^8 PFU/mL were administered every 14 (± 3) days for up to approximately 9 months.
  Talimogene laherparepvec was administered by intralesional injection only into injectable cutaneous, subcutaneous, nodal tumors, and other non-visceral tumors with or without image ultrasound guidance.
Period: Overall Study
Arm/Group | Cohort A1: Talimogene Laherparepvec (TVEC) - Aged 12 to ≤ 21 Years | Cohort B1: Talimogene Laherparepvec (TVEC) - Aged 2 to < 12 Years
Started | 13 | 2
Received Talimogene Laherparepvec | 13 | 2
Completed | 0 | 0
Not Completed | 13 | 2
Not completed — Death | 12 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A1: Talimogene Laherparepvec (TVEC) - Aged 12 to ≤ 21 Years | Cohort B1: Talimogene Laherparepvec (TVEC) - Aged 2 to < 12 Years | Total
Number analyzed (Participants) | 13 | 2 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.2 (2.8) | 9.0 (2.8) | 14.3 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 8 | 2 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 10 | 1 | 11
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 2 | 11
  Other | 3 | 0 | 3
  American Indian or Alaska Native | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced a Dose-limiting Toxicity (DLT)
Description: All toxicities were graded using the Common Terminology Criteria for Adverse Events version 4.0:
  * Grade 1: Mild
  * Grade 2: Moderate
  * Grade 3: Severe/medically significant but not immediately life-threatening
  * Grade 4: Life-threatening
  * Grade 5: Death related to adverse event
  The occurrence of any of the below was considered a DLT, if judged to be related to talimogene laherparepvec:
  * Grade 4 non-hematologic toxicity
  * Grade 3 non-hematologic toxicity that lasted > 3 days despite optimal supportive care
  * Any ≥ grade 3 non-hematologic laboratory value if medical intervention was required, the abnormality led to hospitalization or the abnormality persisted for > 1 week unless deemed not clinically important per both investigator & sponsor
  * Febrile neutropenia grade 3/4
  * Thrombocytopenia < 25 x 10^9/L associated with bleeding event that required intervention
  * Serious herpetic event
  * Grade 5 toxicity
  * Any intolerable toxicity that led to permanent discontinuation of talimogene laherparepvec
Time Frame: Day 1 to Day 35
Population: DLT Analysis Set: all DLT evaluable participants defined as participants who had the opportunity to be followed for at least 35 days from the initial dosing of talimogene laherparepvec and received at least two treatments of talimogene laherparepvec (except participants who had a DLT after the first dose).
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Cohort A1: Talimogene Laherparepvec (TVEC) - Aged 12 to ≤ 21 Years | Cohort B1: Talimogene Laherparepvec (TVEC) - Aged 2 to < 12 Years
Number analyzed (Participants) | 11 | 2
Percent of participants
  Experienced a DLT | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 84.2]
  Did Not Experience a DLT | 100.0 [71.5 to 100.0] | 100.0 [15.8 to 100.0]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who experienced either complete response (CR) or partial response (PR) per modified immune-related response criteria simulating Response Evaluation Criteria in Solid Tumors (irRC-RECIST) response criteria.
  CR was defined as the disappearance of all lesions (whether measurable or not and whether baseline or new) and confirmation by a repeat, consecutive assessment no less than 4 weeks (28 days) from the date first documented. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR was defined as the decrease in tumor burdena ≥ 30% relative to baseline confirmed by a consecutive assessment at least 4 weeks (28 days) after first documentation.
Time Frame: Every 12 weeks until the end of follow-up; maximum duration of follow-up was 54.51 months
Population: Safety Analysis Set: all participants who received at least one dose of talimogene laherparepvec.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A1: Talimogene Laherparepvec (TVEC) - Aged 12 to ≤ 21 Years | Cohort B1: Talimogene Laherparepvec (TVEC) - Aged 2 to < 12 Years
Number analyzed (Participants) | 13 | 2
Percentage of participants | 0.0 [0.00 to 24.71] | 0.0 [0.00 to 84.19]

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the date of an initial response of CR or PR to the earlier of PD/death.
Time Frame: Every 12 weeks until the end of follow-up; maximum duration of follow-up was 54.51 months
Population: Safety Analysis Set: all participants who received at least one dose of talimogene laherparepvec.
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort A1: Talimogene Laherparepvec (TVEC) - Aged 12 to ≤ 21 Years | Cohort B1: Talimogene Laherparepvec (TVEC) - Aged 2 to < 12 Years
Number analyzed (Participants) | 13 | 2
Days | NA [NA to NA] — No participants experienced a response of CR or PR, so DOR could not be calculated. | NA [NA to NA] — No participants experienced a response of CR or PR, so DOR could not be calculated.

4. Secondary Outcome: Time to Response (TTR)
Description: TTR was defined as the number of days from the first dose of talimogene laherparepvec to the first objective assessment of response as per modified irRC-RECIST.
Time Frame: Every 12 weeks until the end of follow-up; maximum duration of follow-up was 54.51 months
Population: Safety Analysis Set: all participants who received at least one dose of talimogene laherparepvec.
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort A1: Talimogene Laherparepvec (TVEC) - Aged 12 to ≤ 21 Years | Cohort B1: Talimogene Laherparepvec (TVEC) - Aged 2 to < 12 Years
Number analyzed (Participants) | 13 | 2
Days | NA [NA to NA] — No participants experienced a response of CR or PR, so TTR could not be calculated. | NA [NA to NA] — No participants experienced a response of CR or PR, so TTR could not be calculated.

5. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time from the first dose of talimogene laherparepvec until objective tumor progression per irRC-RECIST.
  TTP was estimated using the Kaplan-Meier method.
Time Frame: Every 12 weeks until the end of follow-up; maximum duration of follow-up was 54.51 months
Population: Safety analysis set: all participants who received at least one dose of talimogene laherparepvec.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A1: Talimogene Laherparepvec (TVEC) - Aged 12 to ≤ 21 Years | Cohort B1: Talimogene Laherparepvec (TVEC) - Aged 2 to < 12 Years
Number analyzed (Participants) | 13 | 2
Months | 2.50 [0.00 to 9.0] | NA [1.6 to 3.5] — Insufficient participants experienced disease progression, so the median could not be calculated.

6. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the first dose to the earlier of disease progression per modified irRC-RECIST or death from any cause.
  PFS was estimated using the Kaplan-Meier method.
Time Frame: Every 12 weeks until the end of follow-up; maximum duration of follow-up was 54.51 months
Population: Safety analysis set: all participants who received at least one dose of talimogene laherparepvec.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A1: Talimogene Laherparepvec (TVEC) - Aged 12 to ≤ 21 Years | Cohort B1: Talimogene Laherparepvec (TVEC) - Aged 2 to < 12 Years
Number analyzed (Participants) | 13 | 2
Months | 3.32 [1.1 to 11.6] | 6.42 [1.6 to 11.2]

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as as the time from first dose to the event of death from any cause.
  OS was estimated using the Kaplan-Meier method.
Time Frame: Every 12 weeks until the end of follow-up; maximum duration of follow-up was 54.51 months
Population: Safety Analysis Set: all participants who received at least one dose of talimogene laherparepvec.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A1: Talimogene Laherparepvec (TVEC) - Aged 12 to ≤ 21 Years | Cohort B1: Talimogene Laherparepvec (TVEC) - Aged 2 to < 12 Years
Number analyzed (Participants) | 13 | 2
Months | 9.40 [1.1 to 54.5] | 8.02 [4.8 to 11.2]

ADVERSE EVENTS:
Time Frame: Mortality: Day 1 until end of follow-up; The median [min, max] duration of follow-up was 9.396 [1.12, 54.51] months Adverse events: From first dose of study drug until 30 days after last dose. The median [min, max] duration of treatment was 1.18 [0.0, 9.1] months in T-VEC Cohort A1 and 2.81 [2.0, 3.6] months in T-VEC Cohort B1
Description: Adverse events and serious adverse event are reported for all participants who received at least one dose of talimogene laherparepvec. Duration of treatment = ((The date of last dose of study drug - The date of first dose of study drug + 1)/365.25 * 12).
Arm/Group | Cohort A1: Talimogene Laherparepvec (TVEC) - Aged 12 to ≤ 21 Years | Cohort B1: Talimogene Laherparepvec (TVEC) - Aged 2 to < 12 Years
All-Cause Mortality (participants affected / at risk) | 12/13 | 2/2
Serious Adverse Events (participants affected / at risk) | 5/13 | 1/2
Other Adverse Events (participants affected / at risk) | 13/13 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A1: Talimogene Laherparepvec (TVEC) - Aged 12 to ≤ 21 Years (N=13) | Cohort B1: Talimogene Laherparepvec (TVEC) - Aged 2 to < 12 Years (N=2)
Nausea (Gastrointestinal disorders) | 1 | 0
Vascular device infection (Infections and infestations) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Osteosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cranial nerve disorder (Nervous system disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A1: Talimogene Laherparepvec (TVEC) - Aged 12 to ≤ 21 Years (N=13) | Cohort B1: Talimogene Laherparepvec (TVEC) - Aged 2 to < 12 Years (N=2)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Autoimmune hypothyroidism (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 6 | 1
Asthenia (General disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Face oedema (General disorders) | 1 | 0
Fatigue (General disorders) | 4 | 0
Influenza like illness (General disorders) | 3 | 0
Injection site inflammation (General disorders) | 1 | 0
Injection site pain (General disorders) | 2 | 0
Malaise (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 0
Pyrexia (General disorders) | 9 | 2
Drug hypersensitivity (Immune system disorders) | 1 | 0
Influenza (Infections and infestations) | 2 | 0
Mastitis (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Heat cramps (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1
Headache (Nervous system disorders) | 5 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 0
Presyncope (Nervous system disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Disease progression (General disorders) | 1 | 1
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
General physical condition abnormal (Investigations) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Participant recruitment ended when 15 participants were enrolled due to difficulties in enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT02756845/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT02756845/SAP_001.pdf